CLINICAL TRIAL: NCT01342458
Title: Therapeutic Effect of Inexpensive, Flexible and Non-heeled Footwear on the Clinical, Functional and Gait Biomechanics in Elderly Women With Knee Osteoarthritis: a Randomized Clinical Trial
Brief Title: Effect of Footwear on the Clinical, Functional, and Biomechanical Aspects in Elderly Women With Knee Osteoarthritis (OA)
Acronym: OA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Francis Trombini, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LABIMPH_OA2
Record Dates: First submitted 2011-04-20; First posted 2011-04-27 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Shoes; Gait; Biomechanics
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Daily use of the intervention Flexible footwear (Moleca®) for 6 months, for at least 42 hours/week (approximately 6 hours/day, 7 days/week). The Moleca® shoe (Calçados Beira Rio S.A., Novo Hamburgo, Rio Grande do Sul, Brazil) is a low-cost women's double canvas, flexible, flat, walking shoe without heels, with a 5-mm anti-slip rubber sole and a 3-mm flat insole of ethylene vinyl acetate that provides only protection but no correction. The mean weight of the shoe is 0.172±0.019 kg (range 0.091 to 0.182 kg), depending on size. This minimalist footwear is commonly worn by the elderly of all social classes and its average cost is US$ 6.25.
  Interventions: Other: Flexible footwear
- Control Group (No Intervention): During the intervention period, patients from the Control Group (CG) were instructed not to wear Flexible footwear (Moleca®) or other similar minimalist footwear. During everyday activities, the CG group was only permitted to wear a standard, neutral tennis shoe. At the end of the intervention period, all CG participants also received one pair of Moleca® shoes at no cost.

INTERVENTIONS:
Other: Flexible footwear — The patients of the Intervention Group (IG) will be use over 6 month a flexible and non-heeled footwear (Moleca; Calçados Beira Rio S.A., Novo Hamburgo, Rio Grande do Sul, Brazil) is a women's flexible flat walking shoe, without heels, with an anti-slip rubber sole, 5-mm thin, with a 3 mm internal wedge of ethylene vinyl acetate, made out of dubbed canvas. It had a mean weight of 172 ± 19.6 g, ranging from 142 to 193 g depending upon the size.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to determine whether inexpensive, flexible and non-heeled footwear is effective in improving of clinical, functional and gait biomechanics in elderly women with knee osteoarthritis.

DETAILED DESCRIPTION:
* The clinical and functional aspects will be evaluated using a visual analogue scale (VAS) for pain, Western Ontario and McMaster Universities (WOMAC) and Lequesne questionnaires of quality of life in patients with knee osteoarthritis and testing of six-minute walk (6MWT).
* Biomechanical analysis of gait will be performed by infrared cameras and a force platform. From the data of kinematics and kinetics, will be calculated moments of the knee joint strength by inverse dynamics.

The process (steps) will be divided as follows:

* step 1, in this step there will be sorting and initial assessment of potential participants; pain will be evaluated through VAS, function and quality of life by means of questionnaires WOMAC and Lequesne and the 6MWT, and by evaluating the biomechanics of gait.
* step 2,(3 month follow-up), both groups will be evaluated again by the VAS and WOMAC and Lequesne questionnaires.
* step 3, after 6 months of starting the monitoring process, both groups will be reevaluated through the VAS, WOMAC, Lequesne, 6MWT and biomechanical analysis of gait. This step is the final evaluation, characterizing the end of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Kellgren and Lawrence grade 2 or 3
* Being able to walk independently for at least 6 hours per day without the aid of canes or attendant to perform their activities of daily living
* Knee pain between 3 and 8 on the visual analogue scale

Exclusion Criteria:

* Previous history of surgery on knees, ankles and hips in the last 2 years
* Neurological disease
* BMI > 35 kg/m2
* Difference in lower limb length > 1 cm
* Prostheses and / or lower limb orthoses
* Having received steroid injections and hyaluronic acid intra-articular knee in previous periods of three and six months respectively
* Present at the knee joint instability (positive test results in the medial collateral ligament, lateral, anterior and posterior drawer)
* OA of the hip and / or ankle incapacitating or diagnosed OA in lower limbs and spine
* Inflammatory arthritis (eg. rheumatoid arthritis)
* Asymptomatic OA of one or both knees
* Dementia or inability to provide consistent information
* Introduction of Nonsteroidal Anti-inflammatory Drugs and analgesic medications 8 weeks before inclusion or change of dosage of the same after the inclusion
* Being under physiotherapy or acupuncture treatment
* Patients with an indication of prosthesis or orthosis
* Patients who are already using a flexible and non-heeled shoes for more than 25 hours per week (3 ½ hours per day) over the past 6 months

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel CN Sacco, PhD, Principal Investigator — Department of Physical therapy, Speech, and Occupational Therapy, School of Medicine, University of Sao Paulo
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Trombini-Souza F, Fuller R, Goldenstein-Schainberg C, Sacco ICN. Long-term use of minimal footwear in older adult women with knee osteoarthritis: Mechanisms of action in the knee adduction moment. J Biomech. 2020 Jul 17;108:109885. doi: 10.1016/j.jbiomech.2020.109885. Epub 2020 Jun 13. PMID 32635999
- [Derived] Trombini-Souza F, Matias AB, Yokota M, Butugan MK, Goldenstein-Schainberg C, Fuller R, Sacco IC. Long-term use of minimal footwear on pain, self-reported function, analgesic intake, and joint loading in elderly women with knee osteoarthritis: A randomized controlled trial. Clin Biomech (Bristol). 2015 Dec;30(10):1194-201. doi: 10.1016/j.clinbiomech.2015.08.004. Epub 2015 Aug 14. PMID 26307181
- [Derived] Trombini-Souza F, Fuller R, Matias A, Yokota M, Butugan M, Goldenstein-Schainberg C, Sacco IC. Effectiveness of a long-term use of a minimalist footwear versus habitual shoe on pain, function and mechanical loads in knee osteoarthritis: a randomized controlled trial. BMC Musculoskelet Disord. 2012 Jul 12;13:121. doi: 10.1186/1471-2474-13-121. PMID 22788574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited from the primary care centre of the School of Medicine, University of São Paulo Hospital, and rheumatology ambulatory medical. Participants were recruited between March 2011 and December 2012, and allocated equally into one of two groups.
Groups:
- Intervention Group: Daily use of the intervention footwear (Moleca®) for 6 months, for at least 42 hours/week (approximately 6 hours/day, 7 days/week). The Moleca® shoe (Calçados Beira Rio S.A., Novo Hamburgo, Rio Grande do Sul, Brazil) is a low-cost women's double canvas, flexible, flat, walking shoe without heels, with a 5-mm anti-slip rubber sole and a 3-mm flat insole of ethylene vinyl acetate that provides only protection but no correction. The mean weight of the shoe is 0.172±0.019 kg (range 0.091 to 0.182 kg), depending on size. This minimalist footwear is commonly worn by the elderly of all social classes and its average cost is US$ 6.25.
- Control Group: During the intervention period, patients from the Control Group (CG) were instructed not to wear Moleca® or other similar minimalist footwear. During everyday activities, the CG group was only permitted to wear a standard, neutral tennis shoe. At the end of the intervention period, all CG participants also received one pair of Moleca® shoes at no cost.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 28 | 28
Completed | 26 | 24
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Population: Tests t were used to provide similar characteristics between the both groups for the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (5) | 66 (6) | 66 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities (WOMAC) Pain Subscale
Description: The WOMAC (Western Ontario and McMaster Universities) pain subscale consists of five questions (Likert Scale) relating to the patient's pain in everyday situations. The Likert Scale version used for all WOMAC items are: none, mild, moderate, severe, and extreme. The sum of all items of pain subscale ranges from 0 to 20. Higher scores indicate worse pain.
Time Frame: 6 month
Population: An intention-to-treat analysis was performed, and the missing data were treated as missing completely at random (MCAR) using the Mahalanobis imputation method (SOLAS software version 4.0; Statistical Solutions Ltd., Cork, Ireland).
Measure: Mean (Standard Deviation); unit: score
Groups:
- Intervention Group; Control Group: WOMAC pain subscale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 26 | 24
score
  WOMAC pain (Baseline) | 9.2 (4.0) | 10.0 (3.9)
  WOMAC pain (3rd month) | 4.5 (2.3) | 6.6 (4.7)
  WOMAC pain (6th month) | 3.1 (2.2) | 7.2 (4.8)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Sample size was calculated based on pain WOMAC score and was accomplished using a moderate effect size (f=0.30). Standard deviation estimates were taken from our previous study. A sample size of 56 patients was needed to provide 80% power for detecting a moderate effect difference between the highest and lowest group pain means, with an alpha level of 0.05, a statistical design of F test of repeated measures (between and within effects), and assuming a 10% loss to follow-up; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intervention Group; From baseline to 3rd month; Test type: Superiority or Other; p < 0.001, post hoc newman keuls; Effect Size = 1.46
Statistical Analysis 3: Comparison: Intervention Group; From baseline to 6th month; Test type: Superiority or Other; p < 0.001, post hoc Newman Keuls; Effect size = 1.94
Statistical Analysis 4: Comparison: Control Group; From baseline to 3rd month; Test type: Superiority or Other; p = 0.001, post hoc Newman-Keuls; Effect size = 0.82
Statistical Analysis 5: Comparison: Control Group; From baseline to 6th month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.66

2. Secondary Outcome: WOMAC Stiffness Subscale
Description: The stiffness subscale included in the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) index consists of two questions (Likert Scale) relating articular function of the patient. The Likert Scale version used for all WOMAC items are: none, mild, moderate, severe, and extreme. The sum of all items of the stiffness subscale ranges from 0 to 8. Higher scores on the stiffness WOMAC subscale indicate worse articular function.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score
Groups:
- Intervention Group; Control Group: WOMAC stiffness subscale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 26 | 24
score
  WOMAC Stiffness subscale (Baseline) | 1.8 (1.9) | 2.4 (2.3)
  WOMAC Stiffness subscale (3rd month) | 0.8 (0.9) | 2.9 (2.1)
  WOMAC Stiffness subscale (6th month) | 0.7 (1.1) | 2.0 (2.4)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; We used a casewise two-way ANOVA for repeated measures (two independent groups and three repeated measures/assessments), followed by a post hoc Newman-Keuls to verify the interaction effect of group vs. time between T0 (baseline), T3 (3th month) and T6 (6th month); Test type: Superiority or Other; p = 0.015, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intervention Group; From baseline to 3rd month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.66
Statistical Analysis 3: Comparison: Intervention Group; From baseline to 6th month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.70
Statistical Analysis 4: Comparison: Control Group; From baseline to 3rd month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.25
Statistical Analysis 5: Comparison: Control Group; From baseline to 6th month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.16

3. Secondary Outcome: WOMAC Physical Function Subscale
Description: The physical function subscale included in the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) index consists of seventeen questions (Likert Scale) relating to the patient's physical activities, or skills to move out and take care of themselves. The Likert Scale version used for all WOMAC items are: none, mild, moderate, severe, and extreme. The sum of all items of physical function subscale ranges from 0 to 68. Higher scores on the physical function WOMAC subscale indicate worse functional limitations.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score
Groups:
- Intervention Group; Control Group: WOMAC Physical function subscale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 26 | 24
score
  WOMAC Physical function subscale (Baseline) | 27.6 (14.3) | 29.6 (13.2)
  WOMAC Physical function subscale (3rd month) | 13.2 (7.3) | 20.9 (12.8)
  WOMAC Physical function subscale (6 month) | 10.2 (6.5) | 23.9 (14.8)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; We used a casewise two-way ANOVA for repeated measures (two independent groups and three repeated measures/assessments), followed by a post hoc Newman-Keuls test to verify the interaction effect of group vs. time between T0 (baseline), T3 (3th month) and T6 (6th month); Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intervention Group; From baseline to 3rd month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 1.28
Statistical Analysis 3: Comparison: Intervention Group; From baseline to 6th month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 1.58
Statistical Analysis 4: Comparison: Control Group; From baseline to 3rd month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.68
Statistical Analysis 5: Comparison: Control Group; From baseline to 6th month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.42

4. Secondary Outcome: WOMAC Total Score
Description: The WOMAC total score is the sum of all subscale (pain, function and stiffness) (Likert Scale) relating to the patient's physical activities, or skills to move out and take care of themselves. The Likert Scale version used for all WOMAC items are: none, mild, moderate, severe, and extreme. The sum of all items ranges from 0 to 96. Higher scores on the WOMAC total score indicate worse condition.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score
Groups:
- Intervention Group; Control Group: The WOMAC total score is the sum of all subscale (pain, function and stiffness).
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 26 | 24
score
  WOMAC total score (Baseline) | 37.7 (17.9) | 42.0 (17.3)
  WOMAC total score (3rd month) | 17.6 (8.9) | 30.4 (18.3)
  WOMAC total score (6th month) | 14.3 (8.8) | 33.8 (20.3)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intervention Group; From baseline to 3rd month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 1.45
Statistical Analysis 3: Comparison: Intervention Group; From baseline to 6th month; Test type: Superiority or Other; p = 0.019, post hoc Newman-Keuls; Effect size = 1.69
Statistical Analysis 4: Comparison: Control Group; From baseline to 3rd month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.66
Statistical Analysis 5: Comparison: Control Group; From baseline to 6th month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.44

5. Secondary Outcome: Global Score of the Lequesne´s Questionaire Algo-functional.
Description: This questionaire consists of three sections (eleven questions): about pain or discomfort, the maximum distance that the patient can walk, and activities of daily living. Scores range from zero to twenty-four, meaning cases without involvement and with extremely severe impairment, respectively.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score
Groups:
- Intervention Group; Control Group: Global score of the Lequesne´s questionaire algo-functional.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 26 | 24
score
  Lequesne (Baseline) | 9.7 (3.5) | 11.5 (3.3)
  Lequesne (3rd month) | 6.3 (3.1) | 8.9 (4.3)
  Lequesne (6th month) | 5.5 (3.2) | 9.7 (4.7)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intervention Group; From baseline to 3rd month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 1.07
Statistical Analysis 3: Comparison: Intervention Group; From baseline to 6th month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 1.31
Statistical Analysis 4: Comparison: Control Group; From baseline to 3rd month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.71
Statistical Analysis 5: Comparison: Control Group; From baseline to 6th month; Test type: Superiority or Other; p < 0.001, post hoc Newman-Keuls; Effect size = 0.45

6. Secondary Outcome: Six-minute Walk Test
Description: The six-minute walk test assesses distance in meters walked over 6 minutes.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: meter
Groups:
- Intervention Group; Control Group: Six-minute walk test
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 26 | 24
meter
  Six-minute walk test (Baseline) | 433.5 (48.9) | 430.6 (56.8)
  Six-minute walk test (3rd month) | 453.5 (40.6) | 431.6 (43.1)
  Six-minute walk test (6th month) | 439.3 (34.7) | 428.3 (44.2)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.425, Mixed Models Analysis

7. Secondary Outcome: First Peak of the Knee Adduction Moment (KAM) During Gait.
Description: The first peak of the external knee moment was calculated by mean inverse dynamics approach. To this procedure, we used the kinematics data of the lower limbs assessed with six infrared cameras and the ground reaction force evaluated by mean a force platform. This is a continuous measure.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: % body weight x height in centimeters
Groups:
- Intervention Group; Control Group: Knee adduction moment (KAM) first peak
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 26 | 24
% body weight x height in centimeters
  KAM (Baseline) | 2.44 (0.77) | 2.21 (1.06)
  KAM (6th month) | 2.37 (0.63) | 2.28 (1.12)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.443, Mixed Models Analysis

8. Secondary Outcome: Paracetamol Intake
Description: Paracetamol intake (500 mg), number of tablets per month.
Time Frame: 6 month
Measure: Median (Inter-Quartile Range); unit: tablets per month
Groups:
- Intervention Group; Control Group: A rescue analgesic medication (paracetamol) was allowed only if necessary (2g/day max.)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 26 | 24
tablets per month | 0 [0 to 3] | 10 [6 to 24]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Difference in paracetamol intake at 6-month; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 10

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 1/28 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=28) | Control Group (N=28)
Keratosis on metatarsal head (Musculoskeletal and connective tissue disorders) | 1 | 0 — Keratosis on the head of the fifth metatarsal in left foot .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No